CLINICAL TRIAL: NCT04904237
Title: Azacytidine-venetoclax Combination as Leukemia Debulking Treatment Followed by Reduced Toxicity Conditioning Regimen (Melphalan Busulfan and Fludarabine, MBF) as Salvage Therapy for Refractory Acute Myeloid Leukemia (AML).
Brief Title: Aza-Ven Followed by Reduced Toxicity Conditioning Regimen (MBF) as Salvage Therapy for Refractory AML.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head BMT program, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-rAML-2021
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Refractory Acute Myeloid Leukemia
Keywords: refractory; acute myeloid leukemia; hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aza-ven +MBF (Experimental): treatment with aza-ven debulking therapy followed by allo-HSCT with MBF conditioning
  Interventions: Drug: Aza-Ven-allo-HSCT

INTERVENTIONS:
Drug: Aza-Ven-allo-HSCT — aaa-ven treatment followed by allo-HCTS with reduced toxicity conditioning (RTC) of Fludarabine, Busulifan and Melphalan
  Other Names: Aza-Ven MBF

SUMMARY:
In this phase clinical trail, we evaluate the efficacy and feasibility of azacytidine and venetoclax as leukemia debulking treatment followed by reduced intensity conditioning regimen consisting of Fludarabine + Busulfan + Melphalan as salvage treatment in patients with refractory AML .

DETAILED DESCRIPTION:
In refractory AML, allogeneic hematopoietic stem cell transplantation (allo-HCST) is considered as the only curative regimen. In this phase II clinical trial, we plan to evaluate the efficacy and feasibility of new sequential transplantation protocol. All patients receive azacytidine and venetoclax as leukemia debulking treatment which is followed by reduced intensity conditioning regimen consisting of Fludarabine (150mg/m2) + Busulfan (6.4mg/kg) + Melphalan (70mg/m2). The graft-versus host disease (GVHD) prophylaxis regimen is based on reduced dose of post-transplantation cyclophosphamide (PT-CY) 40mg/kg day+3~+4, tacrolimus and low-dose anti-thymoglobulin (ATG, 2.5mg/kg) in case of HLA-matched unrelated donor or halo-donor transplantation.

ELIGIBILITY:
Inclusion Criteria:

* refractory AML (no remission after 2 induction therapy, relapsed AML within 6 months of first complete remission (CR), relapse AML no CR after reinduction therapy), multiple relapse and refractory relapse AML
* patients with HLA matched related or unrelated donor (9~10/10) or haplo-identical related donor

Exclusion Criteria:

* Patients with poor liver function (enzyme >2N or bilirubin >2N)
* poor renal function (Scr >1.5N)
* poor cardiac function （EF<45%）
* inform consent not provided

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival | 12 months
  event defined as relapse or death of any causes

SECONDARY OUTCOMES:
overall survival | 12 months
  event defined as death of all causes
non-relapse mortality | 12 months
  event defined as death of all causes other than leukemia relapse
relapse | 12 months
  event defined as leukemia relapse
GVHD and relapse free survival (GRFS) | 12 months
  event defined as leukemia relapse, death of any causes, III-IV aGVHD or moderate to severe cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, Principal Investigator — Shanghai Rui Jin Hospital
Locations (3):
- China (3):
  - Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai
  - Department of Hematology, Shanghai No6 Hospital, Shanghai
  - Shanghai ZhaXin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No